CLINICAL TRIAL: NCT07187479
Title: Randomized, Open Label Study to Examine the Outcomes of Physiologic Insulin Resensitization in Patients With Chronic Kidney Disease and Type 2 Diabetes Mellitus
Brief Title: Outcomes of Physiologic Insulin Resensitization (PIR) in Patients With Chronic Kidney Disease and Type 2 Diabetes Mellitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Well Cell Global (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZ-01
Record Dates: First submitted 2025-09-18; First posted 2025-09-23 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Chronic Kidney Disease (Stages 4 and 5); Kidney Disease; Type 2 Diabetes
Keywords: chronic kidney disease; type 2 diabetes; diabetes; kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Randomized, Open Label Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physiologic Insulin Resensitization (PIR) Group (Experimental): Subject to receive Physiologic Insulin Resensitization (PIR)
  Interventions: Other: Physiologic Insulin Resensitization (PIR)
- Standard of Care (SOC) Group (No Intervention): Subjects will receive standard of care

INTERVENTIONS:
Other: Physiologic Insulin Resensitization (PIR) — PIR is a physician-directed treatment that uses an exterior infusion pump to deliver insulin intravenously.
  Arms: Physiologic Insulin Resensitization (PIR) Group

SUMMARY:
The purpose of this research is to evaluate outcomes of physiologic insulin re-sensitization (PIR) in patients with Chronic Kidney Disease (CKD) and Type 2 Diabetes Mellitus (T2DM).

DETAILED DESCRIPTION:
The primary objective of this study is to assess the outcomes of Physiologic Insulin Resensitization (PIR) treatment compared to standard of care (SOC) on renal patients with a diagnosis of chronic kidney disease (CKD) (stages 3b, 4 and 5) and Type 2 diabetes mellitus (T2DM)

ELIGIBILITY:
Inclusion Criteria:

* Is age 18 or older (male or female)
* Have a documented diagnosis of CKD stage 3b, 4, or 5 and T2DM of 6 months or greater prior to screening. Patients may have treatment regimens associated with T2DM that include diabetic oral and/or injectable medications including insulin and/or GLP-1 receptor agonists.
* In the opinion of the Investigator, has been on an appropriate, stable regimen for management of any complications present for the past six (6) months.
* In the opinion of the Investigator, is able to do all of the following:

  * Provide valid informed consent.
  * Understand and comply with study procedures as presented in the consent process.
  * Has the capacity or support to attend all required visits.
* If female, the subject must meet either of the following sets of conditions:

  o Is of non-childbearing potential, defined as meeting either of the following criteria:
* Age ≥50 years and post-menopausal for at least one (1) year
* Surgically sterile due to bilateral tubal ligation, bilateral oophorectomy, or hysterectomy
* Is of childbearing potential and meets both of the following criteria:

  * Has a negative serum pregnancy test (beta-human chorionic gonadotropin) at screening.
  * Agrees to practice an acceptable method of birth control (contraception) from screening until at least 30 days after last study treatment

Exclusion Criteria:

* Has in the past two (2) years received treatment for a malignancy.
* Current pregnancy or intends to become pregnant during the study
* Has in the past one (1) year used non-prescription opioids or psychoactive drugs.
* Has in the past six (6) months had a hypoglycemic event requiring urgent care and/or administration of glucagon, osteocalcin, or parenteral glucose, unless approved for enrollment by the Medical Monitor.
* Has within the past one (1) month participated in a clinical study involving either of the following:

  * An investigational drug or procedure for any clinical indication
  * An investigation method for glucose control using approved agents
* Is nursing or is planning to nurse during the study.
* Has at screening a positive test for HIV (4th gen. screen), HBsAg, or HCV viral load.
* Has at screening, one or more of the following abnormal lab results:

  * Hb <8 g/dL
  * WBC <2,000/µL
  * Platelets <50,000/µL
  * ALT, AST, or Alkaline Phosphatase >5x ULN
  * ALT or AST >2.5x ULN, and Total Bilirubin >2x ULN
  * Serum albumin <3 g/dL
* Has - in the opinion of the Investigator - psychiatric, behavioral, cognitive and/or clinical dysfunction (whether or not related to known medical illness or drug / alcohol use) that would affect the subject's safety and/or compliance.
* Is on active dialysis at time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Estimated Glomular Filtration Rate (eGFR) | 12 and 24 weeks
  Assess the eGFR of patients in the PIR group as compared to the SOC group
Blood Urea Nitrogen/Creatinine Ratio (BUN/Cr) | 12 and 24 weeks
  Assess the BUN/Cr of patients in the PIR group as compared to the SOC group
Cystatin C | 12 and 24 weeks
  Assess the Cystatin C of patients in the PIR group as compared to the SOC group
Urine albumin-creatinine ratio (ACR) | 12 and 24 weeks
  Assess the urine ACR of patients in the PIR group as compared to the SOC group

SECONDARY OUTCOMES:
Prescribed medication usage for control of symptoms | 12 and 24 weeks
  Assess changes of medications in the PIR group as compared to the SOC group
Hemoglobin A1c (HbA1c) | 12 and 24 weeks
  Assess the Hb1c of patients in the PIR group as compared to the SOC group
Fasting blood glucose | 12 and 24 weeks
  Assess the fasting blood glucose of patients in the PIR group as compared to the SOC group
Fasting insulin level | 12 and 24 weeks
  Assess the fasting insulin level of patients in the PIR group as compared to the SOC group
HOMA-IR | 12 and 24 weeks
  Assess the HOMA-IR of patients in the PIR group as compared to the SOC group
Blood Pressure | 12 and 24 weeks
  Assess the Blood Pressure of patients in the PIR group as compared to the SOC group
Lipid profile | 12 and 24 weeks
  Assess the Lipid Profile of patients in the PIR group as compared to the SOC group
C peptide | 12 and 24 weeks
  Assess the C peptide of patients in the PIR group as compared to the SOC group
EQ-5D-5L Quality of Life (EuroQol 5-Dimension 5-Level Questionnaire) | 12 and 24 weeks
  Assess the Quality of Life of patients in the PIR group as compared to the SOC group. Lower health index scores reflect greater health deficits.

CONTACTS AND LOCATIONS:
Overall Officials: Sungchun Lee, MD, Principal Investigator — Arizona Kidney Disease and Hypertension Centers
Locations (1):
- Arizona Kidney Disease and Hypertension Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing plan is to be determined.